CLINICAL TRIAL: NCT02149082
Title: Near-infrared Spectroscopy (NIRS) for Intracranial Hematoma Detection in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 14-010812
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Intracranial Hematoma
Keywords: Intracranial hematoma; traumatic brain injury; Near infrared spectroscopy; NIRS
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Infrascanner exam: Infrascanner Model 2000 exams may be conducted either before or after an associated head CT for pediatric patients presenting to the emergency department (ED) or pediatric intensive care unit (PICU) with a known or suspected traumatic head injury undergoing a head CT scan to evaluate for the presence or absence of an intracranial hematoma. The time between the head CT scan and the Infrascanner exam will be within 6 hours. The exam involves placing a sensor on the designated areas of the head with the most common locations for traumatic hematoma. Readings from the monitor evaluating each region will be evaluated and recorded. The 8-point exam can be accomplished within 5 minutes or less.
  Interventions: Device: Infrascanner Model 2000

INTERVENTIONS:
Device: Infrascanner Model 2000 — The Infrascanner Model 2000 device is a small, portable handheld device that uses near infrared (NIR) technology to screen patients for intracranial bleeding.

SUMMARY:
This is a study to determine whether the Near infrared spectroscopy (NIRS) optical density (OD) measurement with an Infrascanner device accurately identifies the presence of an intracranial hematoma in pediatric patients ≤18 years of age after known or suspected traumatic brain injury compared with head computerized tomography (CT) scans as the gold standard.

DETAILED DESCRIPTION:
A key decision point in the management of patients with an acute traumatic brain injury is determining the presence of an intracranial hematoma that may require neurosurgical intervention. An expanding hematoma can lead to significant neurological morbidity or death due to brainstem compression or further ischemic injury. Unfortunately, no single physical sign, symptom, or score reliably indicates the presence of an intracranial hematoma. A computerized tomography (CT) scan of the head is the gold standard for emergent identification and localization of acute intracranial hematomas. However, the ionizing radiation from CT scans is associated with an increased risk of developing malignancies. Near infrared spectroscopy (NIRS) is a non-invasive technology that may be useful as an adjunctive modality to CT scanning for early identification of intracranial hematomas. A hand-held NIRS device called the Infrascanner has shown about 90% sensitivity and specificity for detecting intracranial hematomas in adults and a few small studies have shown similar results in children. The present study will aim to validate this device in a wide age range of pediatric subjects and in multiple hospital settings where this device may serve as a valuable screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≤18 years admitted to the Children's Hospital of Philadelphia (CHOP) ED or PICU with a known or suspected traumatic head injury undergoing a head CT scan to evaluate for the presence of an intracranial hematoma.
* Head injury occurred <12 hours prior to presentation for the initial CT scan, or the subject had a clinical change prompting repeat CT scanning.

Exclusion Criteria:

* Evidence of extensive scalp injury including lacerations, avulsions, or abrasions that will impair proper coupling of the Infrascanner device to the subject's head or prevent placement of the device in the specified locations.
* History of neurosurgical procedure (e.g. decompressive craniectomy) with residual bone flap.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Emergency Department (ED), Pediatric Intensive Care Unit (PICU)
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2014-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity of NIRS Optical Density (OD) Measurement | 2-years
  Determine the sensitivity of the NIRS optical density measurement by the Infrascanner device for identifying the presence of intracranial hematomas in pediatric patients after known or suspected traumatic brain injury compared to head CT scans as the gold standard

SECONDARY OUTCOMES:
Specificity and Predictive Values of NIRS Measurement | 2-years
  Determine the specificity, as well as positive and negative predictive values of the NIRS measurement for detecting intracranial hematomas
Variability in Sensitivity and Specificity Based on Hematoma Characteristics | 2-years
  Determine whether sensitivity and specificity vary depending on hematoma type (i.e. epidural, subdural, subarachnoid, intracerebral), hematoma volume, distance of hematoma from brain surface, and skull thickness
Age Varying Sensitivity | 2-years
  Determine whether the sensitivity of the NIRS measurement differs by patient age.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kirschen, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States